CLINICAL TRIAL: NCT03963414
Title: A Phase I Study of Durvalumab (MEDI4736) Plus Tremelimumab in Combination With Platinum-based Chemotherapy in Untreated Extensive-Stage Small Cell Lung Cancer and Performance Status 2
Brief Title: A Study of Durvalumab Plus Tremelimumab With Chemotherapy in Untreated ES-SCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Nebraska (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0275-19-FB
Record Dates: First submitted 2019-04-29; First posted 2019-05-24 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Extensive stage small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; tremelimumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Durvalumab 1500 mg via IV infusion every 3 weeks, starting on Week 7, for up to a maximum of 2 doses/cycles followed by durvalumab maintenance monotherapy 1500 mg via IV infusion every 4 weeks, starting 4 weeks after Cycle 4.
  Interventions: Combination Product: Durvalumab in combination with carboplatin and etoposide
- Cohort 2 (Experimental): Durvalumab 1500 mg plus tremelimumab 75 mg via IV infusion every 3 weeks, starting on Week 7, for up to a maximum of 2 doses/cycles followed by durvalumab monotherapy 1500 mg via IV infusion every 4 weeks, starting 4 weeks after the last infusion of the combination.
  Interventions: Combination Product: Durvalumab + Tremelimumab in combination with carboplatin and etoposide

INTERVENTIONS:
Combination Product: Durvalumab + Tremelimumab in combination with carboplatin and etoposide — 1500mg of durvalumab plus 75mg of tremelimumab in combination with carboplatin and etoposide will be given every 3 weeks for Cycles 3 and 4. 1500mg of durvalumab plus 75mg of tremelimumab will be given every 3 weeks for Cycles 5 and 6.
  Other Names: MEDI4736
  Arms: Cohort 2
Combination Product: Durvalumab in combination with carboplatin and etoposide — 1500mg of durvalumab in combination with carboplatin and etoposide will be given every 3 weeks for Cycles 3 and 4.
  Other Names: MEDI4736
  Arms: Cohort 1

SUMMARY:
This study is designed to evaluate the safety and tolerability of durvalumab and tremelimumab in combination with intravenous (IV) carboplatin plus (+) etoposide in new patients with extensive-stage small cell lung cancer (ES-SCLC).

DETAILED DESCRIPTION:
This Phase I, multicenter, study is designed to evaluate the safety and tolerability of durvalumab (anti-programmed death-ligand 1 [PD-L1] antibody) and tremelimumab (anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4] antibody) in combination with intravenous (IV) carboplatin plus (+) etoposide in treatment naïve patients with extensive-stage small cell lung cancer (ES-SCLC) and performance status 2 (PS2). Eighteen patients with untreated ES-SCLC and PS2 will be enrolled. Cohort 1, which includes the first 6 subjects, will receive IV carboplatin and etoposide Q 3 weeks x 4 cycles. Durvalumab 1500 mg IV Q 3 weeks will be given with chemotherapy during cycles 3 and 4. This will be followed by durvalumab 1500 mg IV Q 4 weeks until disease progression. If 2 out of 6 patients have dose-limiting toxicities, then the study will be closed. Cohort 2, which will include 12 additional subjects, will receive chemotherapy Q 3 weeks x 4 cycles. Durvalumab 1500 mg IV + tremelimumab 75 mg IV Q 3 weeks will be given with chemotherapy during cycles 3 and 4, then durvalumab 1500 mg + tremelimumab 75 mg will be administered Q 3 weeks during cycles 5 and 6. This will be followed by durvalumab 1500 mg IV Q 4 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at time of study entry (consent) and adult male or female (For Nebraska, ≥19 years old)
2. Histologically or cytologically confirmed ES-SCLC
3. Tumor biopsy or cytology should be obtained within 8 weeks of initiation of treatment.
4. Brain metastases; must be asymptomatic or treated and stable, off steroids for at least 1 month prior to study treatment.
5. Have not received any prior therapy for SCLC, except palliative radiation. If the patient received radiation, there must be measurable disease outside the radiation field.
6. Measurable disease or evaluable disease based on RECIST Version 1.1.
7. Eastern Cooperative Oncology Group ECOG = 2
8. Body weight > 30 kg
9. No active secondary malignancy. Patients with other prior malignancies will be included, provided they have been disease-free for at least five years.
10. Adequate hematologic and end organ function
11. Women of childbearing potential must have a pregnancy test (urine or serum) proven negative within 14 days prior to registration.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 28 days.
2. Any previous chemotherapy and /or immunotherapy for SCLC
3. Current or prior use (≤ 14 days before first doses of study drugs) of immunosuppressive medication.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
5. History of another primary malignancy except for malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP
6. History of leptomeningeal carcinomatosis
7. Paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic steroids or clinical symptomatology suggesting worsening of PNS
8. Active infection including tuberculosis, HIV, hepatitis B and C.
9. Active or prior documented autoimmune or inflammatory disorders
10. Uncontrolled cardiovascular disease
11. History of active primary immunodeficiency
12. Pregnant or lactating women
13. Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events with a Severity of 3 or higher (Safety and tolerability) | 3 months
  Evaluate the safety and tolerability profile of durvalumab + tremelimumab in combination with carboplatin and etoposide in ES-SCLC and PS2. Adverse events with a severity grade of 3 or higher per CTCAE guidelines will be used to assess this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Apar Ganti, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No